CLINICAL TRIAL: NCT01253980
Title: The Efficacy of Prophylactic Antibiotics in the Management of Pneumonitis Following Paraffin (Kerosene) Ingestion in Children
Brief Title: Antibiotic Efficacy in Pneumonitis Following Paraffin (Kerosene) Ingestion in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Kate Balme, Dr, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 095/2010; PACTR201201000259370 (Registry Identifier: Pan African Clinical Trial Registry)
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Results first posted 2013-06-26 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-10

CONDITIONS: Kerosene Pneumonitis
Keywords: pneumonitis; paraffin; kerosene
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxicillin (Active Comparator): Amoxicillin
  Interventions: Drug: Amoxicillin
- Placebo suspension (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin — Amoxicillin syrup 20-30mg/kg 8 hourly for 5 days
  Arms: Amoxicillin
Drug: Placebo — Placebo suspension made of water, dextrose and glycerine with a similar taste and appearance to the active comparator.
  Dose 20-30mg/kg 8 hourly for 5 days
  Arms: Placebo suspension

SUMMARY:
Paraffin (kerosene) ingestion in the developing world accounts for a large number of visits to healthcare facilities, especially amongst children. There is no evidence in animals and no good evidence in humans that the use of early antibiotics improves the clinical outcome of paraffin-induced pneumonitis. This randomised placebo-controlled trial will investigate whether the use of early antibiotics affects the clinical course of children with pneumonitis following paraffin ingestion.

DETAILED DESCRIPTION:
The average of 100 children per annum attending Red Cross War Memorial Children's Hospital 9RCWMCH) with the diagnosis of kerosene ingestion would give a sample of 200 children over a two-year period, with 100 patients in each group. From a postulated secondary infection rate of 15 to 50% for children not receiving an antibiotic, a midway point of 25% estimated the treatment failure rate in the placebo group. With no information available on the treatment failure rate in the active group, failure rates of 10% and 5% were arbitrarily applied. With 25% and 5% treatment failure rates for placebo and active groups respectively, at a level of significance of α = 0.05 a sample size of 100 per group gives a power of 0.98 and with failure rates of 25% and 10% a power of 0.80.

Statistical analysis was done using IBM SPSS Version 20 (SPSS Inc., Chicago, IL, USA). Categorical variables are expressed as n (%) and continuous variables as median (interquartile range (IQR)). A P value of ≤ 0.05 was considered significant for all situations. For categorical variables, Fischer's exact test was used for small samples or less frequent occurrences. Chi-Square testing was applied for larger samples or more frequent occurrences. Mann-Whitney or Kruskal-Wallis tests were used for ordinal and continuous variables. Significant correlation between factors and covariates (Spearman's rank coefficient) favoured univariate analysis over binary logistic regression modelling to determine potential risk factors for treatment failure. Continuous variables were categorised for clinical relevance or logistic regression testing. In some instances, specific clinical parameters or reported symptoms were not recorded or the presence or absence of a risk factor was unknown. The missing values, unknown factors and the flow of patient follow-up account for totals not always adding up to the full number of study participants. In the results for Day 3 and Day 5 post-ingestion, the denominator used to calculate proportions for reported symptoms included those patients who attended and who were telephone interviewed, whereas the denominator for clinical signs was only the patients who attended.

The primary outcome measure was treatment failure, as reported. Secondary outcome measures were length of hospital stay, reported symptoms (cough, shortness of breath, wheeze and fever) and clinical signs (respiratory rate, flaring, recessions, grunting, wheeze, crepitations, temperature and altered mental status) at follow-up at Day 3 and 5 post-ingestion for placebo and active groups. Further investigation explored the role of confounding conditions (upper respiratory tract infection, active Mycobacterium tuberculosis infection) and risk factors for treatment failure or delayed resolution (vomiting post-ingestion, household smoking contact, HIV exposure status, prior respiratory history, young age etc). Secondary outcome measures, confounding conditions and risk factors are not reported in this Clinical Trials format, but are reported in the PI's Master's thesis. (Balme KH. The efficacy of prophylactic antibiotics in the management of pneumonitis following paraffin (kerosene) ingestion in children [Master's thesis]. [Cape Town]: University of Cape Town; 2013. 113 p.)

ELIGIBILITY:
Inclusion Criteria:

* Ingestion in the preceding 24 hours
* Presence of respiratory symptoms and/or signs at presentation
* Informed consent obtained from parent or legal guardian
* Resident within the Red Cross Hospital drainage area and able to come for two follow-up appointments

Exclusion Criteria:

* Asymptomatic and no clinical signs
* Too ill to be excluded from receiving an antibiotic as judged by:

  * Requiring more than 2L/min nasal-prong oxygen
  * Requiring continuous or intermittent positive airway pressure ventilation
  * Fever > 40˚C
* Needing an antibiotic for another reason e.g. otitis media, tonsillitis
* Current antibiotic use, prior to kerosene ingestion
* Allergic to amoxicillin

Ages: 3 Months to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Zar, MBBCh PhD, Study Director — University of Cape Town; Michael D Mann, MMed Paed PhD, Study Director — University of Cape Town
Locations (1):
- Red Cross War Memorial Children's Hospital, Cape Town, Western Cape, South Africa

REFERENCES:
- [Result] Balme KH, Zar H, Swift DK, Mann MD. The efficacy of prophylactic antibiotics in the management of children with kerosene-associated pneumonitis: a double-blind randomised controlled trial. Clin Toxicol (Phila). 2015;53(8):789-96. doi: 10.3109/15563650.2015.1059943. Epub 2015 Jun 26. PMID 26114347

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 21 July 2010 - 21 September 2011 (24 hours a day) Patients recruited from Medical Emergency Department
Groups:
- Placebo: Placebo 20-30mg per kg 8 hourly for 5 days
- Amoxicillin: Amoxicillin 20-30mg per kg 8 hourly for 5 days
Period: Overall Study
Arm/Group | Placebo | Amoxicillin
Started | 35 | 39
Completed | 35 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Amoxicillin | Total
Number analyzed (Participants) | 35 | 39 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 39 | 74
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 19 [15 to 21] | 20 [16 to 24] | 19 [16 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 21 | 24 | 45
Region of Enrollment [Number; unit: participants]
  South Africa | 35 | 39 | 74

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: A treatment failure was a patient who at any time deteriorated necessitating a change to the treatment regimen. This was determined by assessing reported symptoms (cough, shortness of breath, wheeze and fever) and comparing clinical signs (respiratory rate, oxygen saturation, wheeze, flaring, grunting, recessions, crepitations, temperature, mental status) to signs at presentation.
Time Frame: At routine follow-up 3 and 5 days post-ingestion or earlier if necessary
Population: per protocol
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Placebo | Amoxicillin
Number analyzed (Participants) | 35 | 39
participants | 3 [3 to 22] | 2 [1 to 17]
Statistical Analysis 1: Comparison: Placebo vs Amoxicillin; Test type: Superiority or Other; p > 0.50, Fisher Exact; Relative risk = 0.60, 95% CI 2-sided [0.11 to 3.37]

ADVERSE EVENTS:
Time Frame: 5 days
Description: The study was not testing a new drug, but rather reviewing efficacy of a known drug compared to placebo. Drug was not given to children with known allergy to amoxicillin. There were no idiosyncratic drug reactions. No children had events which could be linked to the study drug; any clinical findings were related to the kerosene pneumonitis.
Arm/Group | Placebo | Amoxicillin
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/39
Other Adverse Events (participants affected / at risk) | 0/35 | 0/39

LIMITATIONS AND CAVEATS:
Early termination leading to small number of participants. Some patients did not attend follow-up and were only contacted by phone, therefore clinical data not available for all participants at follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No